CLINICAL TRIAL: NCT06687564
Title: Role of ACTG2 Variants in Smooth Muscle Determination and Function in Pediatric Intestinal Pseudo-obstruction.
Acronym: SMOOTH-PIPO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC23.0368; 2024-A01516-41 (Other: ID RCB)
Record Dates: First submitted 2024-10-11; First posted 2024-11-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: PIPO
Keywords: PIPO; CIPO; ACTG2; pseudo-obstruction; organoid; iPS; Pediatric Intestinal Pseudo-Obstruction; Chronic Intestinal Pseudo-obstruction
MeSH Terms: conditions — Intestinal Pseudo-Obstruction | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Experimental, descriptive, prospective, non-randomized, controlled, comparative, monocentric in recruitment but multicentric study in procedures and analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIPO patients (Experimental): PIPO patients with variants of interest
  Interventions: Procedure: Biopsy
- WT (Other): Control arm, same experiments as for patients. Samples from specific cell lines
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — A skin biopsy and a blood sample will be taken to culture the iPS cells and intestinal organoids.
  Other Names: Blood sample

SUMMARY:
The primary objective of this study is to describe the transcriptional impact of R178, R257, R40 or A136 variants of the ACTG2 gene on iPS differentiation mechanisms up to organoids derived from PIPO patient samples versus those derived from control / WT patients (generation of IPS from cultured cell lines), at different stages of their experimental ex vivo development.

DETAILED DESCRIPTION:
Recruited patients will be sampled during a consultation: a blood sample and a biopsy will be taken directly from the patient. Once these samples have been taken, they will be cultured to be reprogrammed into iPS cells, then grown and differentiated into intestinal organoids.

Various experiments will be carried out (as described in the outcomes) to identify at molecular, cellular and tissue level the mechanisms altered in patients with an R178, R257, R40 or A136 variant, assessing their consequence(s) on the development and functionality of the digestive mesenchyme.

ELIGIBILITY:
Inclusion Criteria:

PIPO Population:

1. Minor or adult patient ≥ 4 years of age
2. Patient with PIPO before age 18
3. Male or female
4. Patient with PIPO meeting at least 2 of the ESPGHAN criteria (Thapar et al 2018) and carrying the R178, R257, R40 or A136 mutation of the ACTG2 gene.
5. Patient whose assent has been obtained and whose legal guardians have given their written informed consent
6. Patient affiliated to the French Social Security system or benefiting from an equivalent plan

WT population:

- iPS cell lines MS573 or WT8288 or 202CT or SD378M, from the Nantes University Hospital biological collection and generated from samples from control patients without POIC who have consented to donate their samples.

Exclusion Criteria:

PIPO population :

1. Patients with a history of radiotherapy treatment
2. Patient with lymphocyte lineage damage

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Description of the transcriptional impact of R178, R257, R40 or A136 variants of the ACTG2 gene | At different stages of their experimental ex vivo development (mesenchymal progenitors, determined smooth muscle cells, differentiated smooth muscle cells and 3D organization of smooth muscle) through study completion, an average of 5 years
  Difference in transcript expression (%) in RNASeq transcriptomic analysis between samples carrying the R178, R257, R40 or A136 variants of the ACTG2 gene on the differentiation mechanisms of iPS up to organoids derived from PIPO patient samples versus those derived from control patients

SECONDARY OUTCOMES:
Evaluate the impact of R178, R257, R40 or A136 variants of the ACTG2 gene on gastrointestinal contractile function between mutant versus WT organoids. | At different stages of their experimental ex vivo development (mesenchymal progenitors, determined smooth muscle cells, differentiated smooth muscle cells and 3D organization of smooth muscle) an average of 5 years
  Difference (%) in isometric contraction force between mutant versus WT organoids by electrical stimulation and specific agonist.
Evaluate the immunofluorescence labeling differential between mutant and WT cells from IPS and organoids | At different stages of their experimental ex vivo development (mesenchymal progenitors, determined smooth muscle cells, differentiated smooth muscle cells and 3D organization of smooth muscle) an average of 5 years
  Difference in fluorescence (%) between mutant and WT cells as cell stages from iPS to organoids
Evaluate the impact of R178, R257, R40 or A136 mutations of the ACTG2 gene on the actin network of fibroblasts derived from skin samples of diseased patients versus those of WTpatients. | At different stages of their experimental ex vivo development (mesenchymal progenitors, determined smooth muscle cells, differentiated smooth muscle cells and 3D organization of smooth muscle) an average of 5 years
  Difference in actin network labeling by immunofluorescence (%) between skin fibroblasts from PIPO and WT patients.
Evaluate the effect of reversion of the R178, R257, R40 or A136 mutation versus WT on functionality and contractility during differentiation of cells into organoids. | At different stages of their experimental ex vivo development (mesenchymal progenitors, determined smooth muscle cells, differentiated smooth muscle cells and 3D organization of smooth muscle) an average of 5 years
  Difference in isometric contraction strength (%) between mutant versus WT versus revertant organoids via specific agonist and electrical stimulation.
Assessing the potential of a chemical library to correct the phenotype | At different stages of their experimental ex vivo development (mesenchymal progenitors, determined smooth muscle cells, differentiated smooth muscle cells and 3D organization of smooth muscle) an average of 5 years
  Identification of molecules inducing a significant difference in isometric contraction force (%) between treated mutant organoids, untreated mutant organoids and treated and untreated WT

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Phymedexp Inserm U1046 - Cnrs Umr 9214, Montpellier
  - Tens - Inserm Un Umr 1235, Nantes
  - AP-HP Hôpital Robert Debré, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zenzeri L, Tambucci R, Quitadamo P, Giorgio V, De Giorgio R, Di Nardo G. Update on chronic intestinal pseudo-obstruction. Curr Opin Gastroenterol. 2020 May;36(3):230-237. doi: 10.1097/MOG.0000000000000630. PMID 32073506
- [Background] Fournier N, Fabre A. Smooth muscle motility disorder phenotypes: A systematic review of cases associated with seven pathogenic genes (ACTG2, MYH11, FLNA, MYLK, RAD21, MYL9 and LMOD1). Intractable Rare Dis Res. 2022 Aug;11(3):113-119. doi: 10.5582/irdr.2022.01060. PMID 36200034
- [Background] Assia Batzir N, Kishor Bhagwat P, Larson A, Coban Akdemir Z, Baglaj M, Bofferding L, Bosanko KB, Bouassida S, Callewaert B, Cannon A, Enchautegui Colon Y, Garnica AD, Harr MH, Heck S, Hurst ACE, Jhangiani SN, Isidor B, Littlejohn RO, Liu P, Magoulas P, Mar Fan H, Marom R, McLean S, Nezarati MM, Nugent KM, Petersen MB, Rocha ML, Roeder E, Smigiel R, Tully I, Weisfeld-Adams J, Wells KO; Baylor-Hopkins Center for Mendelian Genomics; Posey JE, Lupski JR, Beaudet AL, Wangler MF. Recurrent arginine substitutions in the ACTG2 gene are the primary driver of disease burden and severity in visceral myopathy. Hum Mutat. 2020 Mar;41(3):641-654. doi: 10.1002/humu.23960. Epub 2019 Dec 19. PMID 31769566
- [Background] de Santa Barbara P, van den Brink GR, Roberts DJ. Development and differentiation of the intestinal epithelium. Cell Mol Life Sci. 2003 Jul;60(7):1322-32. doi: 10.1007/s00018-003-2289-3. PMID 12943221
- [Background] Mahe MM, Brown NE, Poling HM, Helmrath MA. In Vivo Model of Small Intestine. Methods Mol Biol. 2017;1597:229-245. doi: 10.1007/978-1-4939-6949-4_17. PMID 28361322